CLINICAL TRIAL: NCT03997734
Title: A Phase 1, Placebo-controlled, Randomized, Parallel Group Study to Evaluate the Tolerability, Safety and Pharmacokinetics of a Topical Patch AB001 Following Single and Repeated Administration in Healthy Subjects
Brief Title: Tolerability, Safety and Pharmacokinetics of a Topical AB001 Patch in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABS-102
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Transdermal Patch; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment A-AB001 (Experimental): Apply 1 patch of AB001 patch on the lower back of the subjects on either side of the spine without occlusion for 12 hours on Day 1 in period 1. Subjects who received the AB001 patch in period 1 will then receive a single oral capsule of active ingredient on Day 20 in period 2.
  Interventions: Drug: AB001; Drug: oral capsule
- Treatment B-AB001 (Experimental): Apply 2 patches of AB001 patches on the lower back of the subjects on side of the spine without occlusion for 12 hours on Day 1 and then once daily from Day 8 to 20.
  Interventions: Drug: AB001
- Treatment C (Active Comparator): Apply 1 patch of positive comparative patch on the lower back of the subjects on either side of the spine without occlusion for 48 hours on Day 1 and then one patch every two days from Days 8 to 20.
  Interventions: Drug: positive comparative patch
- Treatment A-Placebo (Placebo Comparator): Apply 1 patch of placebo patch on the lower back of the subjects on either side of the spine without occlusion for 12 hours on Day 1 in period 1.
  Interventions: Drug: Placebos
- Treatment B-Placebo (Placebo Comparator): Apply 2 patches of placebo patches on the lower back of the subjects on side of the spine without occlusion for 12 hours on Day 1 and then once daily from Day 8 to 20.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: AB001 — single and repeated dosing
  Other Names: topical patch
  Arms: Treatment A-AB001; Treatment B-AB001
Drug: oral capsule — single dose
  Other Names: active ingredient
  Arms: Treatment A-AB001
Drug: positive comparative patch — single and repeated dosing
  Other Names: topical patch
  Arms: Treatment C
Drug: Placebos — single and repeated dosing
  Other Names: topical patch
  Arms: Treatment A-Placebo; Treatment B-Placebo

SUMMARY:
The study evaluates the safety, tolerability and pharmacokinetics of single and repeated doses of topical AB001 patch and the bioavailability relative to the oral capsule and topical positive comparative patch.

DETAILED DESCRIPTION:
Eligible subjects will be randomly assigned to Treatment goup A, B and C.

In the experiment group A, 12 subjects with a ratio of 10:2 will receive one patch of AB001 or placebo batch on Day 1 of period 1, respectively, after a wash-out period of 14 days, 10 subjects received AB001 patch will be administered with an oral capsule of active ingredient on Day 20 of period 2.

In the experiment group B, 12 subjects with a ratio of 10:2 will receive two patches of AB001 or two placebo batches on Day 1 respectively, and then two patches daily from Day 8 to Day 20.

In the active comparator group C, 10 subjects will receive one patch of positive comparative patch on Day 1, and then once patch every two days from Day 8 to Day 20.

The tolerability, safety and pharmacokinetics of topical AB001 patch will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between 18 and 45 years with a BMI of 18 to 30 kg/m2, inclusive, and weigh at least 45 kg.
2. Subjects having normal skin without excessive hair growth on tested areas.
3. Evidence of a personally signed and dated informed consent document indicating that the subjects has been informed of all pertinent aspects of the trial.
4. Subjects who are willing to comply with scheduled visits and other trial procedures

Exclusion Criteria:

1. A history or presence of significant cardiovascular, neurological, hematological, psychiatric, infectious, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other conditions known to interfere with the topical absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the investigator
2. History of hypersensitivity to NSAIDs
3. Clinically significant laboratory abnormalities as judged by the investigator
4. Known sensitivity to adhesive tape, component of the test products or topically applied products
5. Any active malignancy
6. Suffering from severe acne, moderate to severe hirsutism or androgenic alopecia
7. Any chronic skin disorder (e.g., eczema, psoriasis) likely to interfere with transdermal drug absorption or assessment of skin tolerability
8. Skin abnormalities likely to be aggravated by the study medication, such as dermatological diseases or infections, rash, skin sensitive to topical preparations or adhesive dressings
9. Pregnant and/or nursing women
10. Any visible skin disorder or abnormal skin pigmentation which, in the opinion of the investigator, would interfere with the outcome of the trial
11. History of alcohol or drug abuse within 18 months
12. Blood donation or significant blood loss within 60 days of dosing or plasma donation within 7 days of dosing
13. Use of any medication within 4 weeks prior to the first treatment or during the trial, which in the opinion of the investigator may influence the trial results or the safety of the subjects
14. Subjects who cannot avoid, throughout the duration of the trial, any swimming, any washing of the back, and sauna or any intense physical activity that might result in excessive sweating
15. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with any adverse events (AEs) | From baseline through Day 26
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of subjects any serious adverse events (SAEs) | From baseline through Day 26
  An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect.

SECONDARY OUTCOMES:
Safety Assessments on Skin Reaction Evaluation | From baseline through Day 26
  Topical Skin Reaction Score(0-2 is a better outcome):
  0= no evidence of irritation
  1. minimal erythema, barely perceptible
  2. definite erythema, readily visible; minimal edema or minimal papular response
  3. erythema and papules
  4. definite edema
  5. erythema, edema and papules
  6. vesicular eruption
  7. strong reaction spreading beyond application site
pharmacokinetic parameters of AB001(Cmax) | Day 1 and Day 26
  Peak Plasma Concentration (Cmax)
pharmacokinetic parameters of AB001 (AUC) | Day 1 and Day 26
  Area under the plasma concentration versus time curve (AUC)
bioavailability of AB001 | Day 1 and Day 26
  To determine the bioavailability of AB001

CONTACTS AND LOCATIONS:
Overall Officials: Frontier clinical team, Study Director — Frontier Biotechnologies Inc.
Locations (1):
- The Third People's Hospital of Wuxi, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No